CLINICAL TRIAL: NCT01244750
Title: Studying Interventions for Managing Patients With Chronic Myeloid Leukemia (CML) in Chronic Phase: The 5-Year Prospective Cohort Study (SIMPLICITY)
Brief Title: Studying First Line Treatment of Chronic Myeloid Leukemia (CML) in a Real-world Setting
Acronym: SIMPLICITY
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CA180-330
Record Dates: First submitted 2010-11-15; First posted 2010-11-19 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Phase - Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- First line TKI treatment: Imatinib: Diagnosed CML patients who receive first line TKI treatment: Imatinib
- First line TKI treatment: Nilotinib: Diagnosed CML patients who receive first line TKI treatment: Nilotinib
- First line TKI treatment: Dasatinib: Diagnosed CML patients who receive first line TKI treatment: Dasatinib
- Imatinib treated patients: Imatinib treated patients if their study index date is between January 2, 2008 and September 30, 2010

SUMMARY:
The purpose of this study is to better understand the use of tyrosine kinase inhibitors (TKI) in patients newly diagnosed with CML and their quality of life in a real-world setting.

DETAILED DESCRIPTION:
Time Perspective : Most patients are expected to be a mix of retrospective and prospective data collection. Patients can be enrolled after their study index date (retrospective component) and have to be followed until 5 years from study index date are complete (time between enrollment and 5 year follow-up is the prospective component)

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed chronic phase chronic myeloid leukemia (CP-CML) patients who started their first-line Tyrosine Kinase Inhibitor (TKI) treatment on imatinib, dasatinib or nilotinib in accordance with the timelines below
* 18 years or older at time of of CP-CML diagnosis

  a) Imatinib Cohorts
* Patients who started their first-line Imatinib treatment between January 2, 2008 and September 30, 2010.Patients fitting this criterion are defined as retrospective Imatinib patients
* Patients who started their first-line Imatinib treatment on or after October 1, 2010

  b) Dasatinib Cohort
* Patients who started their first-line Dasatinib treatment after the drug was approved in this indication

  c) Nilotinib Cohort
* Patients who started their first-line Nilotinib treatment after the drug was approved in this indication
* Patients are also eligible when they have already switched to a subsequent therapy (TKI or other) at the time of enrollment, as long as their first-line and subsequent CML treatment information is available at site for data entry into the study Electronic Case Report Form (eCRF)
* Receiving treatment at medical practice (eg. community-based, office-based, hospital-based, academic setting, oncology center)

Exclusion Criteria:

* Patients who are participating in an interventional trial which may influence the management of their CML disease will be excluded

Discontinuation Criteria:

* Enrolled patients who join an interventional trial which may influence the management of their CML disease will be excluded at the time of entry into the interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at oncology practices or oncology centers linked to a hospital in the North Americas, Europe and potentially at additional sites in South America, and Asia
Sampling Method: Non-Probability Sample
Enrollment: 1494 (Actual)
Dates: Start 2010-12-02 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
The rate of Complete Cytogenetic Response | 12 months
The duration of initial TKI treatment | 5-years from study index date
  Initiation of first-line TKI, (whether Dasatinib, Imatinib, Nilotinib)
The rate of discontinuation and treatment changes after initial TKI treatment | Every 6 months for a follow-up period of 5-years from study index date
  Dates of switches in therapy from initial TKI treatment, Reasons for treatment discontinuation (i.e. side effects, mutations, etc.), Subsequent lines of CML treatments (start and stop dates)
The rate of best response to therapy (i.e. hematologic, cytogenetic, molecular response) | Every 6 months for a follow-up period of 5-years from study index date
  Results and dates of: all bone marrow aspirates, blood tests, cytogenetics, Polymerase Chain Reaction (PCR), Fluorescent In-Situ Hybridization (FISH), and Physical exam
The adherence to treatment | Every 6 months for a follow-up period of 5-years from study index date
  Morisky Medication Adherence Scale - 8 Items is a validated self-reported measure of medication adherence.

SECONDARY OUTCOMES:
Impact of first-line treatment options on quality of life | Every 6 months
  Questionnaires used for assessment:
  Functional Assessment of Cancer Therapy - General (FACT-G), Cancer Therapy Satisfaction Questionnaire (CTSQ), MD Anderson Symptom Inventory - CML (MDASI-CML).
Non-hematologic side effects from treatment affecting patient quality of life and outcomes | Every 6 months
  Treatment discontinuations and changes
Patient satisfaction with CML treatment | Every 6 months
  Cancer Therapy Satisfaction Questionnaire (CTSQ)
Patterns of disease monitoring as observed in a real-world setting | Every 6 months
  MD Anderson Symptom Inventory - CML (MDASI-CML) Questionnaire - disease-specific module of the MDASI7 which is a brief measure of severity and impact of cancer-related symptoms on daily function
Resource utilization associated with CML management | Every 6 months
  To evaluate healthcare resource utilization, descriptive statistics will describe real-world disease monitoring patterns, frequency of testing, and resources used for disease management for each treatment cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (210):
- United States (143):
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC - NAHOA, Sedona, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Little Rock Hematology Oncology Associates, Little Rock, Arkansas
  - Pacific Cancer Medical Center, Inc, Anaheim, California
  - Southwest Cancer Care Medical Group, Escondido, California
  - Wilshire Oncology Medical Group, Inc, Glendora, California
  - University of Southern California, Los Angeles, California
  - St. Joseph's Hospital, Orange, California
  - PMK Medical Group, Inc. DBA Ventura, Oxnard, California
  - Stockton Hematology Oncology, Stockton, California
  - Tahoe Forest Health System Cancer Center, Truckee, California
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Medical Oncology and Blood Disorders, LLP, Manchester, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - Washington Hospital Center, Washington Cancer Institute, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - Hematology And Medical Oncology Of Southern Palm Beach County, Boynton Beach, Florida
  - Broward Oncology Associates, Fort Lauderdale, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Baptist Cancer Institute, Jacksonville, Florida
  - University Of Florida, Jacksonville, Florida
  - Watson Clinic, Lakeland, Florida
  - Central Florida Health Alliance, Leesburg, Florida
  - Baptist Cancer Center, Miami, Florida
  - Florida Cancer Specialists, New Port Richey, Florida
  - Cancer Centers of Florida, Orlando, Florida
  - Lake County Oncology and Hematology, Tavares, Florida
  - Space Coast Cancer Center, Titusville, Florida
  - Peachtree Hematology-Oncology, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Georgia Cancer Specialist, Sandy Springs, Georgia
  - Lewis Hall Singeltary Oncology Center, Thomasville, Georgia
  - OnCare, Honolulu, Hawaii
  - Straub Clinical & Hospital, Honolulu, Hawaii
  - Kaiser Permanente Honolulu, Honolulu, Hawaii
  - Mahafzah Medical Center, Evergreen Park, Illinois
  - Delnor Community Hospital, Geneva, Illinois
  - Mid-Illinois Hem/Onc Asoc, Normal, Illinois
  - North Chicago VA Medical Center, North Chicago, Illinois
  - Southern Illinois School of Medicine, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - Saint John's Cancer Center, Anderson, Indiana
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - Horizon Oncology Research, Inc, Lafayette, Indiana
  - Cancer Care Center, Inc. PC, New Albany, Indiana
  - N. Iowa Mercy Cancer Center, Mason City, Iowa
  - Hutchinson Clinic, Hutchinson, Kansas
  - Cotton O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Louisville Hospital - Brown Cancer Center, Louisville, Kentucky
  - Consultants In Blood Disorders, Saint Matthews, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Willis-Knighton Cancer System, Shreveport, Louisiana
  - Maryland Oncology Hematology Pa, Columbia, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Sturdy Hematology & Oncology Associates, Attleboro, Massachusetts
  - Boston VA Healthcare System, Boston, Massachusetts
  - South Coast Health System, Fall River, Massachusetts
  - Commonwealth Hematology-Oncology, P.C., Quincy, Massachusetts
  - UMass Medical Center, Worcester, Massachusetts
  - Cancer & Hematology Centers of Western Michigan, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Michigan State University, Lansing, Michigan
  - North Mississippi Hematology & Oncology, Tupelo, Mississippi
  - St John's Clinic for Cancer and Hematology, Springfield, Missouri
  - Billings Clinic, Billings, Montana
  - Omaha VAMC, Omaha, Nebraska
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Bms Clinical Research Center, Does Not Exist, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Hematology-Oncology Associates of Northern NJ, PA, Morristown, New Jersey
  - Southern Oncology Hematology, Vineland, New Jersey
  - Broome Oncology, Johnson City, New York
  - Advanced Oncology, New York, New York
  - St. Lukes Roosevelt Medical Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Montefiore Medical Center / AECOM, The Bronx, New York
  - Alamance Regional Cancer Center, Burlington, North Carolina
  - Waverly Hematology Oncology, Cary, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Gaston Hematology Oncology, Gastonia, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Medical Center of Newark, Newark, Ohio
  - Cancer Care Associates, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Hematology/Oncology Salem LLP, Salem, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital and Health Network, Bethlehem, Pennsylvania
  - Medical Oncology Associates of Wyoming Valley, PC, Kingston, Pennsylvania
  - Lancaster General Health, Lancaster, Pennsylvania
  - Veterans Research Foundation of Pittsburgh, Pittsburgh, Pennsylvania
  - Berks Hematology-Oncology, West Reading, Pennsylvania
  - Geisinger Health System, Wilkes-Barre, Pennsylvania
  - Cancer Care Association Of York, York, Pennsylvania
  - Hematology and Oncology Associates of RI, Cranston, Rhode Island
  - The Cancer Center at Memorial Hospital, Pawtucket, Rhode Island
  - Charleston Cancer Center, Charleston, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - Prairie Lakes Healthcare System, Inc, Watertown, South Dakota
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Texas Oncology, Amarillo, Texas
  - Texas Oncology - Arlington South, Arlington, Texas
  - Texas Oncology-Austin North, Austin, Texas
  - Julie & Ben Rogers Cancer Institute, Beaumont, Texas
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Methodist Charlton Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Michael DeBakey VA Medical Center, Houston, Texas
  - Texas Oncology, Lewisville, Texas
  - Texas Oncology-McAllen South Second, McAllen, Texas
  - Texas Oncology, Mesquite, Texas
  - Texas Oncology-Midland Allison Cancer Center, Midland, Texas
  - Texas Oncology-Odessa West Texas Cancer Center, Odessa, Texas
  - Texas Oncology, Paris, Texas
  - North Texas Regional Cancer Center, Plano, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology, Waco, Texas
  - Danville Hematology & Oncology, Danville, Virginia
  - Hematology Oncology Associates of Fredricksburg, Fredericksburg, Virginia
  - Peninsula Cancer Institute, Newport News, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Swedish Cancer Institute-Eastside Hematology/Oncology, Bellevue, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
  - City Hospital - West Virginia University Hospital East, Martinsburg, West Virginia
  - Wheeling Hospital, Wheeling, West Virginia
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
- France (7):
  - Local Institution, Blois
  - Local Institution, Bordeaux
  - Local Institution, Chalon/Saone Cedex
  - Local Institution, Chambéry
  - Local Institution, Le Mans
  - Local Institution, Pierre-Bénite
  - Local Institution, Pringy
- Germany (34):
  - Local Institution, Amberg
  - Local Institution, Aschaffenburg
  - Local Institution, Baden-Baden
  - Local Institution, Bamberg
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Bottrop
  - Local Institution, Coburg
  - Local Institution, Cologne
  - Local Institution, Darmstadt
  - Local Institution, Essen
  - Local Institution, Frankfurt am Main
  - Local Institution, Frankurt Am Main
  - Local Institution, Greifswald
  - Local Institution, Hamm
  - Local Institution, Hof
  - Local Institution, Idar-Oberstein
  - Local Institution, Kaiserslautern
  - Local Institution, Kassel
  - Local Institution, Koblenz
  - Local Institution, Landshut
  - Local Institution, Lebach
  - Local Institution, Leipzig
  - Local Institution, Mülheim A. D. Ruhr
  - Local Institution, Offenbach
  - Local Institution, Potsdam
  - Local Institution, Rostock
  - Local Institution, Rötha
  - Local Institution, Singen
  - Local Institution, Soest
  - Local Institution, Ulm
  - Local Institution, Velbert
  - Local Institution, Weiden
  - Local Institution, Würzburg
- Italy (17):
  - Local Institution, Bari
  - Local Institution, Brescia
  - Local Institution, Brindisi
  - Local Institution, Catania
  - Local Institution, Florence
  - Local Institution, Milan
  - Local Institution, Modena
  - Local Institution, Monza
  - Local Institution, Pavia
  - Local Institution, Perugia
  - Local Institution, Pesaro
  - Local Institution, Rionero in Vulture
  - Local Institution, Roma
  - Local Institution, Rome
  - Local Institution, Siena
  - Local Institution, Terni
  - Local Institution, Udine
- Local Institution, Hoofddorp, Netherlands
- Puerto Rico Hematology Oncology Group, Bayamón, Puerto Rico
- Local Institution, Saint Petersburg, Russia
- Spain (6):
  - Local Institution, Santiago de Compostela-A Coruña, Spain
  - Local Institution, A Coruña
  - Local Institution, Oviedo - Asturias
  - Local Institution, Pamplona
  - Local Institution, Salamanca
  - Local Insitution, Toledo

REFERENCES:
- [Derived] Hehlmann R, Cortes JE, Zyczynski T, Gambacorti-Passerini C, Goldberg SL, Mauro MJ, Michallet M, Simonsson B, Williams LA, Gajavelli S, DeGutis I, Sen GP, Paquette RL. Tyrosine kinase inhibitor interruptions, discontinuations and switching in patients with chronic-phase chronic myeloid leukemia in routine clinical practice: SIMPLICITY. Am J Hematol. 2019 Jan;94(1):46-54. doi: 10.1002/ajh.25306. Epub 2018 Oct 31. PMID 30290003
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Information — http://www.BMSStudyConnect.com